CLINICAL TRIAL: NCT03671278
Title: Implementing the STarT Back Model of Stratifying Care for Patients With Low Back Pain Seeking Care in an Emergency Department: a Prospective Longitudinal Cohort Study
Brief Title: Implementation of the STarT Back Screening Tool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Luciola da Cunha Menezes Costa, Principal Investigator, Universidade Cidade de Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Unicid20
Record Dates: First submitted 2018-09-05; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Low Back Pain
Keywords: low back pain; emergency; feasibility; implementation
MeSH Terms: conditions — Low Back Pain; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STarT Back Screening Tool Approach (Other): After baseline consultation, all patients will receive usual care from their medical doctors as well as an educational booklet and weekly videos containing information on the prognosis of back pain and how patients could deal with their problems. Six weeks after baseline consultation all patients will be screened by the STarT Back Screening Tool (SBST) and will receive a stratified care according to their SBST classification.
  Interventions: Other: STarT Back Screening Tool Approach

INTERVENTIONS:
Other: STarT Back Screening Tool Approach — Patients classified as low risk of persistent pain will be educated about their condition and how to manage their back pain by targeting modifiable prognostic factors. Patients classified as medium risk will receive evidence-based physical therapy. Patients classified as high risk will receive evidence-based physical therapy as well as individualized psychological intervention.

SUMMARY:
The STarT Back Screening Tool (SBST) has been used in different healthcare settings in order to stratify the management of patients with low back pain. However, to date, no study has investigated the feasibility of implementing the SBST in emergency departments. The objective of this study will be to test the implementation of the SBST in the stratification of patients seeking care in emergency departments.

DETAILED DESCRIPTION:
The Start Back Screening Tool (SBST) aims to identify and stratify primary care patients by using modifiable prognostic indicators that are relevant in clinical decision making. The objective of this study will be to test the feasibility of the implementation of the SBST in the stratification of patients seeking care in emergency departments. Study design: A prospective longitudinal cohort study with a 6-month follow-up. Intervention: At 6-weeks after baseline consultation, patients will be targeted to the specific treatment according to their subclassification in the SBST tool: education about pain neurophysiology and physical therapy. This is the first study that will provide results about logistic processes of the implementation of the SBST in the emergency sector, present feasibility data for the conduction of a large randomized controlled trial of subgroups of low back pain.

ELIGIBILITY:
Inclusion Criteria:

* We will include patients with back pain seeking care in emergency departments

Exclusion Criteria:

* We will exclude patients with serious spinal pathologies (such as cancer, fractures, inflammatory and infectious diseases) as well as pregnant patients and patients with nerve root compromise.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility from the perspective of the patient | Adoption at 6 weeks (i.e. at the implementation of treatment after stratification)
  Feasibility will be measured by using 4 constructs (Adoption, adequacy, feasibility and fidelity). These constructs will be measured by using yes/no questions.
Feasibility from the perspective of the patient | Adequacy at 3 months.
  Feasibility will be measured by using 4 constructs (Adoption, adequacy, feasibility and fidelity). These constructs will be measured by using yes/no questions.
Feasibility from the perspective of the patient | Fidelity at 3 months.
  Feasibility will be measured by using 4 constructs (Adoption, adequacy, feasibility and fidelity). These constructs will be measured by using yes/no questions.
Feasibility from the perspective of the patient | Feasibility at 3 months.
  Feasibility will be measured by using 4 constructs (Adoption, adequacy, feasibility and fidelity). These constructs will be measured by using yes/no questions.

SECONDARY OUTCOMES:
Pain intensity measured by a 0-10 Pain Numerical Rating Scale | 1, 2, 6 weeks and 3 and 6 months after first consultation at the emergency department.
  Pain intensity will be measured by an 11-point (0-10) Pain Numerical Rating Scale (Pain NRS). Higher scores indicates higher pain intensity.
Disability measured by the 0-24 Roland Morris Disability Questionnaire | 6 weeks and 3 and 6 months after first consultation at the emergency department.
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire. Higher scores indicates higher disability.
Risk of persistent disability measured by the 0-9 Start Back Screening Tool. | 1, 2, 6 weeks and 3 and 6 months after first consultation at the emergency department.
  Risk of persistent disability will be measured using the 0-9 point Start Back Screening Tool. The higher the score the higher is the risk of persistent disability.
Global Impression of Recovery measured by the -5 to + 5 Global Perceived Effect Scale. | 1, 2, 6 weeks and 3 and 6 months after first consultation at the emergency department.
  Global Impression of Recovery will be measured using the 11-item Global Perceived Effect Scale. Positive values represents recovery and negative values represents deterioration of symptoms.
Recovery from pain | 1, 2, 6 weeks and 3 and 6 months after first consultation at the emergency department.
  Recovery from pain will be measured using a yes/no question (i.e. Were you completely free of back pain over the last month?)
Depressive symptoms over the last week. | 1, 2, 6 weeks and 3 and 6 months after first consultation at the emergency department.
  Depression will be measured by a single question on how depressed patients were over the last week (measured on a 0-10 likert scale)
Recurrence of low back pain symptoms | 6 weeks and 3 and 6 months after first consultation at the emergency department.
  Patients who recovered will be asked if they have experience a recurrence of symptoms

OTHER OUTCOMES:
Out of pocket costs associated with low back pain | 6 weeks and 3 and 6 months after first consultation at the emergency department.
  Out of pocket costs will be measured using a 9-dimension cost diary

CONTACTS AND LOCATIONS:
Overall Officials: Luciola Costa, PhD, Principal Investigator — Universidade Cidade de São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
We can share our dataset upon request.